CLINICAL TRIAL: NCT01858974
Title: Identification of Microbes Through Detection of Pathogen Specific DNA Using Multiplex PCR as a Point of Care Diagnostic Tool in the Setting of Pneumonia
Brief Title: Fast Identification of Pathogen in the Setting of Pneumonia Using Multiplex PCR
Status: Completed | Type: Observational
Sponsor: University of Göttingen (Other)
Collaborators: Curetis AG, Holzgerlingen, Germany (Unknown)
Responsible Party: Principal Investigator, Dr. med. Nils Kunze, Principal Investigator, University of Göttingen
Other Study IDs: ZARI-NK-2013-01
Record Dates: First submitted 2013-05-16; First posted 2013-05-21 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Acute Lower Respiratory Tract Infection; Pneumonia
Keywords: multiplex PCR; MALDI-TOF; pneumonia; microbiological investigation; intensive care
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — aspiration samples from the respiratory system (tracheal secretion sample, BAL) containing microbial DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
With this study the investigators want to determine, if a fast identification of germs, causing infections of the lower respiratory tract, is possible through the use of Multiplex PCR technology - a method that allows on time detection of bacteria in medical specimen by identifying DNA sequences that are known to be specific for the respective microbe. Therefore aspiration samples from the respiratory tracts of ventilated patients, which are suspected to develop such an infection, will be collected and analyzed by using a multiplex PCR (polymerase chain reaction) application situated on the intensive care unit. The investigators want to determine if Multiplex PCR diagnostic could be a faster alternative to conventional microbiological methods. The results of the Multiplex PCR analyses therefore will be compared with results of conventional microbiological methods.

DETAILED DESCRIPTION:
In this clinical observational study it is to be investigated if Multiplex PCR analyses of clinical samples from ventilated critically ill patients could be a fast and accurate alternative to conventional microbiological diagnostic methods in the identification of human pathogenic microbes in the setting of pneumonia. Therefore aspiration samples from intubated and ventilated critically ill patients, which are suspected to develop such an infection, will be collected and analyzed by using a multiplex PCR application situated on the intensive care unit. The samples will be investigated for DNA sequences that are known to be specific for pneumonia causing microbes. Analyses will take place in a point of care setting and will be carried out by intensive care physicians. According to the standard protocols of our intensive care units, conventional microbiological investigations, including MALDI-TOF, will be carried out parallel to the Multiplex PCR analyses.

ELIGIBILITY:
Inclusion Criteria:

* clinical suspicion for an infection of the lower respiratory tract has been raised and decision for microbiological investigation of respiratory aspirate was made

Exclusion Criteria:

* patient has been recruited for a interventional clinical trial
* suspicion for an infection with a germ belonging to risk class 3 and 4 according to the german law (BioStoffV and TRBA, e.g. Mycobacterium tuberculosis)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients will be recruited from two intensive care units of the university hospital.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-06; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Time until pathogen identification through Multiplex PCR | Up to 24 hours after sampling. Sampling (as an iclusion criterion) can be necessary anytime along the ICU stay of the patient (up to 12 months)
  time from sampling until the availability of the results.
time until pathogen identification through conventional microbiological diagnostic methods | Up to 5 days after Sampling. Sampling (as an iclusion criterion) can be necessary anytime along the ICU stay of the patient (up to 12 months).
  time from sampling until the availability of the results.

SECONDARY OUTCOMES:
length of ICU stay | time from ICU admission to ICU discharge of study patients (up to 12 months)
  total LOS ICU
Type and dosage of administered antibiotic therapy | approximately 5 days. Starting with the day the samples are taken. Ending with the day on which the results microbiological test are made avaiable.
  name and dosage of the antibiotic therapeutic agents used to threat the infection

CONTACTS AND LOCATIONS:
Overall Officials: Michael Quintel, Prof. Dr., Study Director — University of Göttingen
Locations (1):
- University Medical Center Göttingen, Göttingen, Lower Saxony, Germany

REFERENCES:
- [Background] Oosterheert JJ, van Loon AM, Schuurman R, Hoepelman AI, Hak E, Thijsen S, Nossent G, Schneider MM, Hustinx WM, Bonten MJ. Impact of rapid detection of viral and atypical bacterial pathogens by real-time polymerase chain reaction for patients with lower respiratory tract infection. Clin Infect Dis. 2005 Nov 15;41(10):1438-44. doi: 10.1086/497134. Epub 2005 Oct 13. PMID 16231254
- [Background] Caliendo AM. Multiplex PCR and emerging technologies for the detection of respiratory pathogens. Clin Infect Dis. 2011 May;52 Suppl 4(Suppl 4):S326-30. doi: 10.1093/cid/cir047. PMID 21460291
- [Derived] Kunze N, Moerer O, Steinmetz N, Schulze MH, Quintel M, Perl T. Point-of-care multiplex PCR promises short turnaround times for microbial testing in hospital-acquired pneumonia--an observational pilot study in critical ill patients. Ann Clin Microbiol Antimicrob. 2015 Jun 13;14:33. doi: 10.1186/s12941-015-0091-3. PMID 26071191